CLINICAL TRIAL: NCT04708665
Title: Iron-deficiency and Non-iron-deficiency Anemia in Pregnancy and Infant Health in India
Brief Title: Iron Deficiency Anemia and Non-iron Deficiency Anemia in Pregnancy in India
Acronym: IDA & NIDA
Status: Completed | Type: Observational
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Lata Medical Research Foundation (Unknown)
Responsible Party: Principal Investigator, Lindsey Locks, Assistant Professor, Boston University Charles River Campus
Other Study IDs: 55207436
Record Dates: First submitted 2021-01-08; First posted 2021-01-14 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Anemia; Anemia, Iron Deficiency; Anemia of Pregnancy
Keywords: Anemia of Pregnancy
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood will be drawn from pregnant women to assess iron status, hemoglobin, and inflammation. Hemoglobin will be assessed with a heel prick in infants and a finger prick in women.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a sub-study nested into the existing NICHD Global Network for Women's & Children's Health Research Maternal Newborn Health (MNH) registry that is a prospective, observational population-based registry in Eastern Maharashtra, India. This study will assess the prevalence of iron deficiency anemia (IDA) and non-iron deficiency anemia (NIDA) in Eastern Maharashtra and will assess the association between both conditions and neo-natal and infant health outcomes (birth weight, gestational age at birth, weight-for-gestational-age z-score and infant hemoglobin concentration at 6 weeks). The investigators will also assess the relative strength of the association between anemia in the 1st trimester and 3rd trimester (after iron needs have increased but mothers may have been taking iron folic acid (IFA) supplements for several months) and infant health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A pregnant women in the first trimester of pregnancy
* Enrolled in the Maternal & Newborn Health Registry
* At least 18 years of age
* Residing in the area of a selected Primary Health Center with the intention to remain in the area through child birth and 6-weeks post-partum

Exclusion Criteria:

* Having multiple fetuses

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 200 pregnant women and their infants in Eastern Maharashtra, India. Mothers will be enrolled in the first trimester of pregnancy and mothers and infants will be followed up until 6 weeks post-partum.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Birthweight | 0-48 hours

SECONDARY OUTCOMES:
gestational age at birth | <48 hours
weight-for-gestational-age z-score | <48 hours
infant hemoglobin at 6 weeks | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey M Locks, ScD MPH, Principal Investigator — Boston University
Locations (1):
- Lata Medical Research Foundation, Nagpur, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No